CLINICAL TRIAL: NCT05597098
Title: Investigation of the Distinct Mechanisms Involved in Inflammatory Resolution Between Healthy Men and Women: RESOLVE-SEX
Brief Title: Investigation of the Distinct Mechanisms Involved in Inflammatory Resolution Between Healthy Men and Women
Acronym: RESOLVE-SEX
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 22/YH/0244
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation | interventions — Cantharidin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Female (Experimental): The participant will initially attend either in person or virtually for a screening visit for eligibility. Cantharidin will be applied on the second visit to the forearm, back or abdomen (depending on patient preference) via 1cm2 cantharidin soaked filter paper. The particpant will then attend for two further cantharidin applications (24 hr and 48 hr after the first application). 72 hours after initial cantharidin application the blister fluid will be collected.
  Interventions: Drug: Cantharidin
- Male (Experimental): The participant will initially attend either in person or virtually for a screening visit for eligibility. Cantharidin will be applied on the second visit to the forearm, back or abdomen (depending on patient preference) via 1cm2 cantharidin soaked filter paper. The particpant will then attend for two further cantharidin applications (24 hr and 48 hr after the first application). 72 hours after initial cantharidin application the blister fluid will be collected.
  Interventions: Drug: Cantharidin

INTERVENTIONS:
Drug: Cantharidin — 0.1% cantharidin solution in acetone from 0.7% stock solution of cantharone is prepared and applied immediately. 10 μl of cantharidin per disc.
  Other Names: Cantharone 0.1%

SUMMARY:
Important differences exist between sexes in incidence, disease patterns and outcomes in coronary artery disease that is not well understood. It is likely that key differences in the underlying biological mechanism, in particular in inflammatory responses, play a part in underpinning these differences. Previous evidence demonstrates that healthy females appear to be more adept at resolving inflammation compared to healthy males. Since inflammation is thought to be a key initiating phenomenon in coronary artery disease the investigators will examine the differences in inflammatory resolution between the sexes in healthy volunteers.

DETAILED DESCRIPTION:
Inflammation is a key process in triggering events caused by coronary artery disease. Indeed, large scale trials have tested the efficacy of a range of anti-inflammatory approaches. However, whilst some of these confirmed the utility of such approaches in leading to reductions in coronary artery disease; the benefits came at a cost with an increased risk of infection. In their previous work the investigators discovered that, women demonstrate enhanced resolution of inflammation compared to males. This accelerated resolution coincided with improved blood vessel function and health. It is also now accepted that a failure of resolution plays an important part in the enhanced inflammation seen in coronary artery disease. Whether the differences in the incidence of coronary artery disease between men and women might be related to differences in their capacity to mount a resolution response is unknown.

To determine whether inflammatory resolution differs between sexes the investigators will use the validated cantharidin-induced model of acute inflammation in healthy volunteers. Previous published studies have shown when cantharidin is applied to the skin it causes acantholysis and blister formation. It is a safe, reproducible technique with no permanent scarring or ill-effects. The investigators will study the effects on inflammatory responses by measuring the levels of cells, inflammatory mediators and markers of vascular function in blister fluid, urine, saliva and blood. Cantharidin application will be applied to separate areas of the skin over the course of three days to create three small blisters in order to examine different timepoints of the inflammatory process. The blister fluid will then be collected on the fourth day which will be analysed according to standard laboratory techniques including flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female volunteers
2. Aged 18-45
3. Volunteers who are willing to sign the consent form

Exclusion Criteria:

1. Healthy subjects unwilling to consent
2. Pregnant, or any possibility that a subject may be pregnant unless in the latter case a pregnancy test is performed with a negative result
3. Current breast feeding
4. History of any serious illnesses, including recent infections or trauma
5. Subjects taking systemic medication (other than the oral contraceptive pill)
6. Subjects with recent (2 weeks) or current antibiotic use
7. Subjects with any history of a blood-borne infectious disease such as Hepatitis B or C virus, or HIV

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2027-12-12 (Estimated); Study Completion 2027-12-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of the presence or not of blister at each timepoint over 24-72h between the sexes | 24 hours, 48 hours, 72 hours
  Visual inspection as to the presence of an intact blister of 24hr, 48 hr and 72 hr cantharidin blisters
Comparison of blister volume at each timepoint over 24-72h between the sexes | 24 hours, 48 hours, 72 hours
  Blister fluid sampled and weighed to determine volume
Comparison of blister cell number at each timepoint over 24-72 hours between the sexes | 24 hours, 48 hours, 72 hours
  Blister fluid collected from 24 hour, 48 hour and 72 hour cantharidin blisters. Fluid will be analysed using standard laboratory techniques including labelled flow cytometry

SECONDARY OUTCOMES:
Comparison of blister leukocyte subsets (neutrophil and monocyte) between the sexes at each timepoint | 24 hours, 48 hours, 72 hours
  Blister fluid collected from 24 hour, 48 hour and 72 hour cantharidin blisters. Fluid will be analysed using standard laboratory techniques including labelled flow cytometry
Comparison of blister lactate levels and LDH between the sexes at each timepoint | 24 hours, 48 hours, 72 hours
  Blister fluid collected from 24 hour, 48 hour and 72 hour cantharidin blisters. Analysis as per standard laboratory techniques.
Comparison of cell death, necrotic, and apoptotic cell numbers between the sexes at each timepoint | 24 hours, 48 hours, 72 hours
  Blister fluid collected from 24 hour, 48 hour and 72 hour cantharidin blisters. Fluid will be analysed using standard laboratory techniques including labelled flow cytometry
4. Comparison of markers of blister efferocytosis between the sexes at each timepoint | 24 hours, 48 hours, 72 hours
  Blister fluid collected from 24 hour, 48 hour and 72 hour cantharidin blisters. Fluid will be analysed using standard laboratory techniques including labelled flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Ahluwalia, BSc PhD, Principal Investigator — Queen Mary University of London
Locations (1):
- The William Harvey Research Institute, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shabbir A, Rathod KS, Khambata RS, Ahluwalia A. Sex Differences in the Inflammatory Response: Pharmacological Opportunities for Therapeutics for Coronary Artery Disease. Annu Rev Pharmacol Toxicol. 2021 Jan 6;61:333-359. doi: 10.1146/annurev-pharmtox-010919-023229. Epub 2020 Oct 9. PMID 33035428
- [Background] Docherty JR, Stanford SC, Panattieri RA, Alexander SPH, Cirino G, George CH, Hoyer D, Izzo AA, Ji Y, Lilley E, Sobey CG, Stanley P, Stefanska B, Stephens G, Teixeira M, Ahluwalia A. Sex: A change in our guidelines to authors to ensure that this is no longer an ignored experimental variable. Br J Pharmacol. 2019 Nov;176(21):4081-4086. doi: 10.1111/bph.14761. Epub 2019 Aug 23. No abstract available. PMID 31441038
- [Result] Rathod KS, Jones DA, Jain AK, Lim P, MacCarthy PA, Rakhit R, Lockie T, Kalra S, Dalby MC, Malik IS, Whitbread M, Firoozi S, Bogle R, Redwood S, Cooper J, Gupta A, Lansky A, Wragg A, Mathur A, Ahluwalia A. The influence of biological age and sex on long-term outcome after percutaneous coronary intervention for ST-elevation myocardial infarction. Am J Cardiovasc Dis. 2021 Oct 25;11(5):659-678. eCollection 2021. PMID 34849299
- [Result] Kapil V, Rathod KS, Khambata RS, Bahra M, Velmurugan S, Purba A, S Watson D, Barnes MR, Wade WG, Ahluwalia A. Sex differences in the nitrate-nitrite-NO* pathway: Role of oral nitrate-reducing bacteria. Free Radic Biol Med. 2018 Oct;126:113-121. doi: 10.1016/j.freeradbiomed.2018.07.010. Epub 2018 Jul 20. PMID 30031863
- [Result] Rathod KS, Kapil V, Velmurugan S, Khambata RS, Siddique U, Khan S, Van Eijl S, Gee LC, Bansal J, Pitrola K, Shaw C, D'Acquisto F, Colas RA, Marelli-Berg F, Dalli J, Ahluwalia A. Accelerated resolution of inflammation underlies sex differences in inflammatory responses in humans. J Clin Invest. 2017 Jan 3;127(1):169-182. doi: 10.1172/JCI89429. Epub 2016 Nov 28. PMID 27893465